CLINICAL TRIAL: NCT04663516
Title: Effectiveness of Exergaming in Reducing Fatigue Among Children With Leukemia
Brief Title: Effectiveness of Exercise Through Video Games in Reducing Fatigue Among Children With Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Afnan Masoud, principle investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ONCO-EXERGAME
Record Dates: First submitted 2020-11-27; First posted 2020-12-11 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Fatigue; Childhood ALL
Keywords: Exergaming; fatigue; Leukemia; Children
MeSH Terms: conditions — Fatigue; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): exercise through video game (Wii)
  Interventions: Other: Exergaming
- control (No Intervention): children in this group will be given advice about the importance of exercising

INTERVENTIONS:
Other: Exergaming — games provided by the console requiring the movement of upper body, lower body and trunk.
  Arms: experimental

SUMMARY:
40 children with cancer who fulfills the inclusion criteria will be included. Participants will be recruited from King Fahad Children's Cancer Center, King Fahad Medical City and King Khaled University Hospital. After obtaining written formal consent, children will be randomly assigned to two groups, control and experimental. Experimental group will play 60 minutes of Wii physical activity games for three weeks, twice each week. while control group will receive conventional therapy. Fatigue will be assessed using pediatric multidimensional fatigue scale- child proxy before, weekly during the study and after. Functional capacity will be measured by six minute walk test before and after study duration, and physical activity will be repeatedly measured by godin-shephard leisure time physical activity questionnaire. All data will be analyzed using appropriate statistical analysis.

DETAILED DESCRIPTION:
The intervention group:

The investigator will:

* handle accompanying each child to the play room, turn on the Wii and ask the child to choose the game he/she prefers to play from the games provided by wii console that requires the movement of the whole body: upper, lower and trunk.
* Monitor the child while playing, helping with the instructions of the game if the child needs assistance as it is only provided in English from the console.
* heart rate and oxygen saturation are planned to be measured every 15 minutes.

The duration is designed to be 60 minutes per session, but the child is allowed to rest for the time needed during the session if he/she feels tired. or if the oxygen saturation of the child reaches 93. or the heart rate reaches the predicted maximum heart rate.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with leukemia, receiving chemotherapy, or off therapy within 6 months.

Exclusion Criteria:

* bone / pulmonary metastasis, having physical or cognitive disability preventing the child from being able to use the controller and board of the console.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
pediatric quality of life multidimensional fatigue scale | one month
  the scale measures fatigue in the dimensions of physical, sleep and rest and cognitive. the validated Arabic version will be used. the total score is 100, the higher the score the better the person is. the lower the score the more fatigued the person is.
six minute walk test | one month
  measures the endurance and capacity of walking, by measuring the distance walked in six minutes of continuous walking. the longer the distance walked in six minutes the better the endurance.

SECONDARY OUTCOMES:
the Godin shepherd leisure time physical activity questionnaire | one week
  measures the units of physical activity done by the child, by multiplying the met value by the minutes of activity done per week. the scale measures units of activity, if one gets 0-18 it means the person is insufficiently active, 18-27 sufficiently active, if more that 27 then the person is active. the questionnaire consists of one question how many days did the person participate in activity, then we should multiply the number of days that person was active by 9 if the activity he/she did was vigorous, by 5 if the activity was moderate and by 3 if the activity was mild.

CONTACTS AND LOCATIONS:
Overall Officials: afnan masoud, Principal Investigator — MSc student
Locations (1):
- King Fahad Medical City, Riyadh, Saudi Arabia